CLINICAL TRIAL: NCT01740856
Title: Randomized Clinical Trial to Assess the Safety of Reducing the Time of Bed Rest Within Five to Three Hours After Diagnostic Cardiac Catheterization With a 6F Sheath
Brief Title: Clinical Trial to Assess the Safety of Reducing the Time of Bed Rest After Cardiac Catheterization
Acronym: Three-Cath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Eneida Rejane Rabelo da Silva, Professor, ScD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS and HCPA 100401
Record Dates: First submitted 2012-10-29; First posted 2012-12-04 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Artery Disease With Myocardial Infarction
Keywords: cardiac catheterization; safety; nursing care; rest; Patients
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1 | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rest three hours (Experimental): Rest three hours
  Interventions: Other: Rest three hours
- Rest five hours (Experimental): Rest five hours
  Interventions: Other: Rest five hours

INTERVENTIONS:
Other: Rest three hours — Intervention group (IG), will maintain bed rest supine for two hours after the digital compression. After this period prescribed, patients sit in bed with the head elevated at 45 degrees for 50 minutes and then walk within the unit hemodynamic for about 10 minutes. Afterwards patients remain sitting out of bed in hemodynamics unit, until they are five hours, then they will be discharge.
  Arms: Rest three hours
Other: Rest five hours — Control group (CG) maintain bed rest supine for four hours after the digital compression. After this period, the patients sit in bed with the head elevated at 45 degrees for 50 minutes and then walk into the unit hemodynamic for 10 minutes. After that patients receive discharge.
  Arms: Rest five hours

SUMMARY:
Reducing the rest time after diagnostic cardiac catheterization for three hours does not increase the complications concerning to the procedure, compared to the rest of five hours.

DETAILED DESCRIPTION:
Reducing the rest time after diagnostic cardiac catheterization for three hours does not increase the complications concerning to the procedure, compared to the rest of five hours. The aim of this study is to compare through a randomized clinical trial to reduce the rest time in bed for five hours after elective diagnostic cardiac catheterization, with a 6F sheath with a transfemoral approach, for a period of three hours of the occurrence of bleeding, hematoma, pseudoaneurysm and a vasovagal reaction.

ELIGIBILITY:
Inclusion Criteria:

* age equal too or above 18 years
* patients undergoing elective diagnostic cardiac catheterization on an outpatient basis and
* who agree to participate by reading and signing the informed consent form.

Exclusion Criteria:

* patients with restriction ambulation;
* users of coumarin anticoagulants;
* IMC greater than 35 kg/m2;
* patients with hypertension (systolic PA > 180 mmHg and diastolic PA > 110 mmHg) at the end of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety | until three days
  Bleeding: seen after the femoral compression after walking and after sitting down ;Hematoma, pseudoaneurysm and bruise: at the site of arterial puncture;vaso-vagal reaction. All of these will be monitoring by telephone contact at 24h, 48h and 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo da Silva, Professor, Principal Investigator — Hospital de Clinicas de Porto Alegre - Graduate Programa from Nursing School at Federal University of Rio Grande do Sul; Roselene Matte, RN, MSc, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil